CLINICAL TRIAL: NCT05173337
Title: Nefopam as a Multimodal Analgesia for Video-assisted Thoracoscopic Surgery
Brief Title: Nefopam as a Multimodal Analgesia for Thoracic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kangbuk Samsung Hospital (Other)
Responsible Party: Principal Investigator, Eunah Cho, MD, Assistant Professor, Kangbuk Samsung Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: NEVATS2
Record Dates: First submitted 2021-08-17; First posted 2021-12-29 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Nefopam

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): Nefopam will not be administered in this group.
- nefopam group (Experimental): Intravenous nefopam 20 mg will be administered twice, immediately after induction of anesthesia and at the end of surgery.
  Interventions: Drug: Nefopam

INTERVENTIONS:
Drug: Nefopam — Nefopam 20 mg is mixed to 100 mL of normal saline, and is infused intravenously over 15 minutes.
  20 mg of nefopam is administered intravenously for two times, after induction and at the end of surgery.
  Arms: nefopam group

SUMMARY:
Acute postoperative pain after video-assisted thoracoscopic surgery is very severe. Because pain after thoracic surgery prevents early recovery, and increases postoperative complications, its is important to prevent pain after video-assisted thoracoscopic surgery. In the present study, we will evaluate whether nefopam reduces pain after video-assisted thoracoscopic surgery.

ELIGIBILITY:
Inclusion Criteria:

* patient scheduled for elective video-assisted thoracoscopic surgery
* American Society of Anesthesiologists physical grade I, II, III
* patient aged from 18 years old

Exclusion Criteria:

* history of allergy in nonsteroidal anti-inflammatory drugs, or nefopam
* renal insufficiency
* liver insufficiency
* myocardial infarction
* glaucoma
* pregnant and lactating women at the time of surgery
* patient who did not consent to the use of patient-controlled analgesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-12-08 (Actual); Primary Completion 2022-09-23 (Actual); Study Completion 2022-09-23 (Actual)

PRIMARY OUTCOMES:
Pain after 1 hour of surgery | 1 hour after surgery.
  Acute postoperative pain will be assessed using numerical rating scale from 0 (no pain) to 10 (worst pain ever).
Pain after 6 hour of surgery | 6 hours hours after surgery.
  Acute postoperative pain will be assessed using numerical rating scale from 0 (no pain) to 10 (worst pain ever).
Pain after 12 hour of surgery | 12 hours after surgery.
  Acute postoperative pain will be assessed using numerical rating scale from 0 (no pain) to 10 (worst pain ever).
Pain after 24 hour of surgery | 24 hours after surgery.
  Acute postoperative pain will be assessed using numerical rating scale from 0 (no pain) to 10 (worst pain ever).

SECONDARY OUTCOMES:
Patient-controlled analgesia use | 24 hours after surgery
  Fentanyl consumption administered thorough the patient-controlled analgesia machine.
Rescue analgesics | 24 hours after surgery.
  Additional analgesic use during postoperative period.

CONTACTS AND LOCATIONS:
Locations (1):
- Eunah Cho, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ki HS, Shim JG, Choi HK, Ryu KH, Kang DY, Park J, Ahn JH, Lee SH, Cho EA. Nefopam as a multimodal analgesia in thoracoscopic surgery: a randomized controlled trial. J Thorac Dis. 2024 Jun 30;16(6):3644-3654. doi: 10.21037/jtd-24-30. Epub 2024 Jun 12. PMID 38983158